CLINICAL TRIAL: NCT05971472
Title: Arthroscopic Repair Versus Opening Wedge High Tibial Osteotomy for Medial Meniscus Posterior Root Tears
Brief Title: Arthroscopic Repair Versus High Tibial Osteotomy for Medial Meniscus Posterior Root Tears
Acronym: Root Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD 169/2021
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Medial Mensical Tear
Keywords: Medial; Meniscus; Posterior; Root; Tear; High Tibial Osteotomy; Arthroscopic Root Repair; Transtibial Pullout; Arthroscopic Repair; Open Wedge
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Who Masked: Participant
Masking Description: single (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic Repair (Active Comparator): Arthroscopic Repair for medial meniscus posterior root tears
  Interventions: Procedure: Arthroscopic Repair
- High tibial osteotomy (Active Comparator): Open wedge High tibial osteotomy for medial meniscus posterior root tears
  Interventions: Procedure: High tibial osteotomy

INTERVENTIONS:
Procedure: Arthroscopic Repair — Arthroscopic Repair for medial meniscus posterior Root tears
  Arms: Arthroscopic Repair
Procedure: High tibial osteotomy — Open Wedge High tibial osteotomy for medial meniscus posterior Root tears
  Arms: High tibial osteotomy

SUMMARY:
The goal of the trial is to compare Arthroscopic repair against Opening wedge high tibial osteotomy for Medial Meniscus posterior root tears

DETAILED DESCRIPTION:
All Patients included in this clinical trial will be informed by written consent will undergo a one week screening to determine the eligibility for study entry.

Patients who meet the eligibility requirements will be randomized in a single blinded manner (patients).

ELIGIBILITY:
Inclusion Criteria:

* Sex: both sexes.
* Age: Above 40
* Degree of Varus: Neutral to 10 degrees of Varus

Exclusion Criteria:

* History of high energy trauma.
* Multiligamentous knee Injury.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Lysholm Score | 3 month and 6 month
  Validated Arabic form of Lyshlom score
IKDC Score | 3 month and 6 month
  Validated Arabic form of IKDC score

SECONDARY OUTCOMES:
infection | 3 month and 6 month
  Occurrence of infection
Non union | 3 month and 6 month
  Occurrence of delayed or non union
Arthrofibrosis | 3 month and 6 month
  Loss of knee ROM or occurrence of Arthrofibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Wael S. Abdel Megid, Professor, Study Director — Ain Shams University; Zeiad M. Zakaria, Assistant Professor, Study Director — Ain Shams University; Radwan G. Abdel Hamid, Assistant Professor, Study Director — Ain Shams University; Mohamed E. Awad, Assistant Professor, Study Director — Ain Shams University
Locations (1):
- Demerdash Hospital, Cairo, Egypt

REFERENCES:
- [Background] Kim KI, Bae JK, Jeon SW, Kim GB. Medial Meniscus Posterior Root Tear Does Not Affect the Outcome of Medial Open-Wedge High Tibial Osteotomy. J Arthroplasty. 2021 Feb;36(2):423-428. doi: 10.1016/j.arth.2020.08.067. Epub 2020 Sep 7. PMID 32978022
- [Background] Nha KW, Lee YS, Hwang DH, Kwon JH, Chae DJ, Park YJ, Kim JI. Second-look arthroscopic findings after open-wedge high tibia osteotomy focusing on the posterior root tears of the medial meniscus. Arthroscopy. 2013 Feb;29(2):226-31. doi: 10.1016/j.arthro.2012.08.027. PMID 23369476
- [Background] Marzo JM, Gurske-DePerio J. Effects of medial meniscus posterior horn avulsion and repair on tibiofemoral contact area and peak contact pressure with clinical implications. Am J Sports Med. 2009 Jan;37(1):124-9. doi: 10.1177/0363546508323254. Epub 2008 Sep 24. PMID 18815238
- [Background] Feucht MJ, Kuhle J, Bode G, Mehl J, Schmal H, Sudkamp NP, Niemeyer P. Arthroscopic Transtibial Pullout Repair for Posterior Medial Meniscus Root Tears: A Systematic Review of Clinical, Radiographic, and Second-Look Arthroscopic Results. Arthroscopy. 2015 Sep;31(9):1808-16. doi: 10.1016/j.arthro.2015.03.022. Epub 2015 May 13. PMID 25979687